CLINICAL TRIAL: NCT02042547
Title: STUDY OF FACTORS FAVORING THE ONSET OF NOVO ATRIAL FIBRILLATION IN THE IMMEDIATE AFTERMATH OF CORONARY ARTERY BYPASS SURGERY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LAURENT PARI 2010
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2010-11

CONDITIONS: Coronary Artery Bypass Graft With or Without ECC
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients about to undergo heart surgery
  Interventions: Other: Tissue samples from the right atrium; Other: Blood samples

INTERVENTIONS:
Other: Tissue samples from the right atrium
Other: Blood samples

SUMMARY:
Before la surgery:

Transthoracic cardiac echography will be done systematically, to measure among other things the size of the left atrium.

During surgery:

Surgery under extracorporeal circulation: tissue samples will be harvested from the right atrium (one before clamping of the aorta (T0= pre-ischemia sample), immediately before declamping of the aorta (T1= post-ischemia sample).

Surgery without extracorporeal circulation: tissue samples from the right atrium before CABG (T0) and a second sample after CABG (T1).

In parallel with the harvesting of cardiac tissue, blood samples will be taken at different times (H0, H3, H24) to correlate tissue data with systemic data. These will be taken by the anesthetists.

After the surgery:

Holter ECG will be set up for 7 days of continuous recording. Each patient will fill in an observation notebook. The biological samples will be analysed immediately and the biological data obtained will be recorded in the observation notebook.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided written informed consent
* Patients covered by the national health insurance scheme
* Heart surgery (CABG) with and without extracorporeal circulation
* Elective or deferred emergency surgery
* Consecutive patients aged less than 80 years

Exclusion Criteria:

* Patients less than 18, under guardianship
* Patients over 18, under guardianship
* Patients who do not understand the study data
* Patients undergoing emergency surgery who therefore cannot be given or understand the explanations for the study (patients in shock, intubated patients with mechanical ventilation)
* History of heart surgery
* History of AF
* Treatment with Cordarone.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary artery bypass graft with or without extracorporeal circulation
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Onset or a de novo episode of atrial fibrillation during the 7 days following heart surgery | 7 days post-surgery

SECONDARY OUTCOMES:
Markers of ischemia: circulating Troponin I before the surgery and at the end of the procedure | Baseline and at the end of surgery (15 minutes after unclamping when extracorporeal circulation)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France